CLINICAL TRIAL: NCT07309159
Title: Impact of Cannabis Consumption on Psychotic Symptoms and Reality Monitoring in Patients With Schizophrenia: a Real-life Study
Acronym: F_r_IEND-3
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Centre Hospitalier Charles Perrens, Bordeaux (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 2025-A01055-44
Record Dates: First submitted 2025-11-24; First posted 2025-12-30 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-11

CONDITIONS: Schizophrenia
Keywords: cannabis; schizophrenia; EMA; reality monitoring
MeSH Terms: conditions — Schizophrenia; Marijuana Abuse | interventions — Ecological Momentary Assessment

STUDY DESIGN:
Intervention Model Description: "Cannabis user" group (SZ-CUD) "Non-cannabis user" group (SZ-noCUD)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- "Cannabis user" group (SZ-CUD) (Experimental): Use of Ecological Momentary Assessment (EMA) and a mobile Reality Monitoring task
  Interventions: Other: Ecological Momentary Assessment (EMA) and Reality Monitoring tasks
- "Non-cannabis user" group (SZ-noCUD) (Active Comparator): Use of Ecological Momentary Assessment (EMA) and a mobile Reality Monitoring task
  Interventions: Other: Ecological Momentary Assessment (EMA) and Reality Monitoring tasks

INTERVENTIONS:
Other: Ecological Momentary Assessment (EMA) and Reality Monitoring tasks — Use of Ecological Momentary Assessment (EMA) and a mobile Reality Monitoring task

SUMMARY:
This study aims to examine the dual effects of cannabis consumption on both positive and negative symptoms of schizophrenia, across laboratory and real-world contexts. By integrating ecological momentary assessment (EMA) with cognitive tasks such as reality monitoring, the research seeks to clarify how cannabis use influences symptom severity and cognitive functioning in individuals with schizophrenia. Gaining insight into these relationships may contribute to the development of more effective management strategies and ultimately improve outcomes for patients living with schizophrenia.

DETAILED DESCRIPTION:
Schizophrenia is a complex psychiatric disorder that affects approximately 1% of the general population, typically emerging in early adulthood. It is characterized by a wide range of symptoms, including positive symptoms (e.g., hallucinations and delusions), negative symptoms (e.g., apathy and emotional blunting), and cognitive impairments. The disorder contributes substantially to the global burden of disease, ranking among the top 30 causes of disability-adjusted life years.

Cannabis use is common among individuals with schizophrenia, with estimates suggesting that between 16% and 42% of patients have used cannabis at some point in their lives. The relationship between cannabis use and schizophrenia is multifactorial. Cannabis consumption has been associated with an increased risk of psychosis, worsening of positive symptoms, and earlier onset of the disorder. However, some studies indicate that cannabis may also exert beneficial effects on negative symptoms, potentially mediated by compounds other than THC.

Cognitive deficits are a core feature of schizophrenia, particularly impairments in reality monitoring. Reality monitoring refers to the ability to distinguish between internally generated events (intrinsic) and those originating from external sources (extrinsic). In schizophrenia, this capacity is often compromised, leading to misattributions of internal thoughts to external sources, which may contribute to the development of positive symptoms such as hallucinations.

Given the dynamic nature of symptoms and substance use in schizophrenia, traditional clinical models may fail to capture the complexity of these interactions. Ecological Momentary Assessment (EMA) provides a novel approach by leveraging mobile devices to collect real-time data on symptoms, substance use, and cognitive performance in everyday life. EMA has been validated in schizophrenia research, offering high-resolution data that can complement and enhance traditional models.

ELIGIBILITY:
Inclusion Criteria:

* DSM-5 diagnosis of schizophrenia or schizo-affective disorder with the following clinical features:

  * Clinically stable and in the residual (non-acute) phase of illness,
  * No change in antipsychotic treatment for at least 1 month,
  * Outpatient, ambulatory care,
  * No uncontrolled positive symptoms (assessed using PANSS)
* Patients able to use a mobile phone.
* Capacity and willingness to give informed consent.
* Must be able to read, speak, and understand French
* Patients subscribing to the French national medical insurance.
* Patients under "curatelle" (partial guardianship) are eligible

Exclusion Criteria:

Patient under "tutelle" (full legal guardianship).

* Psychiatric comorbidities: autism, bipolar disorder.
* Current criteria for any other substance use disorder except for nicotine use disorder.
* Any medical condition hindering the study and/or use of the smartphone application.
* Patients with somatic, cognitive or other disorders preventing the use of the device (deafness, impaired vision, illiteracy….).
* Pregnant or breastfeeding woman.
* Patients who are not proficient in French.
* Subject included in clinical and/or therapeutic experimentation in progress.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Presence of a statistically significant association between cannabis consumption and the reduction of negative symptoms | 8 days
  Presence of a statistically significant association between cannabis consumption and the exacerbation of positive symptoms with EMA scale
Presence of a statistically significant association between cannabis consumption and the exacerbation of positive symptoms | 8 days
  Presence of a statistically significant association between cannabis consumption and the reduction of negative symptoms with EMA scale

CONTACTS AND LOCATIONS:
Overall Officials: David MISDRAHI, MD, Study Director — Centre Hospitalier Charles Perrens

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Argote M, Sescousse G, Brunelin J, Baudin G, Schaub MP, Rabin R, Schnell T, Ringen PA, Andreassen OA, Addington JM, Brambilla P, Delvecchio G, Bechdolf A, Wobrock T, Schneider-Axmann T, Herzig D, Mohr C, Vila-Badia R, Rodie JU, Mallet J, Ricci V, Martinotti G, Knizkova K, Rodriguez M, Cookey J, Tibbo P, Scheffler F, Asmal L, Garcia-Rizo C, Amoretti S, Huber C, Thibeau H, Kline E, Fakra E, Jardri R, Nourredine M, Rolland B. Association between cannabis use and symptom dimensions in schizophrenia spectrum disorders: an individual participant data meta-analysis on 3053 individuals. EClinicalMedicine. 2023 Sep 8;64:102199. doi: 10.1016/j.eclinm.2023.102199. eCollection 2023 Oct. PMID 37731936
- [Result] Addington J, Addington D. Patterns, predictors and impact of substance use in early psychosis: a longitudinal study. Acta Psychiatr Scand. 2007 Apr;115(4):304-9. doi: 10.1111/j.1600-0447.2006.00900.x. PMID 17355521
- [Result] Abdel-Baki A, Lal S, D-Charron O, Stip E, Kara N. Understanding access and use of technology among youth with first-episode psychosis to inform the development of technology-enabled therapeutic interventions. Early Interv Psychiatry. 2017 Feb;11(1):72-76. doi: 10.1111/eip.12250. Epub 2015 May 22. PMID 26011657